CLINICAL TRIAL: NCT01229020
Title: Distribution of Regional Lung Function, as Determined by the Vibration Response Image Generated by the VRI-2000 System as Compared With Standard Radio-nuclear Method
Brief Title: Distribution of Regional Lung Function by Vibration Response Imaging
Status: Completed | Type: Observational
Sponsor: Deep Breeze (Industry)
Responsible Party: Merav Gat / VP of Clinical and Regulatory Affairs, Deep Breeze
Other Study IDs: DB010
Record Dates: First submitted 2010-10-26; First posted 2010-10-27 (Estimated); Last update posted 2010-10-27 (Estimated); Status verified 2010-10

CONDITIONS: Emphysema; COPD
Keywords: Emphysema; COPD; lung sounds; vibration response imaging
MeSH Terms: conditions — Emphysema; Pulmonary Disease, Chronic Obstructive; Respiratory Sounds

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- COPD patients: Patients diagnosed with COPD, by the pulmonologist at the institute,who are referred to undergo ventilation/perfusion scans.
  Interventions: Other: Observational study - no intervention

INTERVENTIONS:
Other: Observational study - no intervention — Observational study - no intervention. Patients underwent VRI recordings and routine V/Q scan.

SUMMARY:
Assessment of regional contribution of different areas of the lung to its integrated function is often required, such as prior to lung resection in the presence of tumor or emphysema. This assessment is derived from the proportion of zonal radionuclear perfusion or ventilation. The investigators hypothesized that lung VRI may provide an alternative approach to assess regional lung function.

DETAILED DESCRIPTION:
Patients diagnosed with moderate-to-severe COPD by lung function studies and clinical evaluation presented in stable clinical condition and were evaluated by lung sound recordings and quantitative V/Q lung scintigraphy. Regional signals (percentage of lung sounds) for left and right lungs were compared with the corresponding regional count percentages of each radionuclide scan, by V/Q scan regions of interest.

ELIGIBILITY:
Inclusion Criteria:

* Patient is able to read and understand the Informed Consent Form and he/she will provide written Informed Consent.
* Male or female in the age range of 18-85 years.
* The patient will undergo V/Q scan (up to ONE WEEK from the VRI recording)
* The patient presented for evaluation of COPD.
* Body Mass Index >21.

Exclusion Criteria:

* Unstable clinical status such as fever, acute shortness of breath, cough, hemoptysis, cheat pain, or acute chest illness.
* Chest wall deformation;
* Spine deformation (including severe scoliosis);
* Hirsutism;
* Potentially contagious skin lesion on the back;
* Skin lesion that would interfere with sensor placement;
* Any additional chronic lung disease of any findings such as past tuberculosis, visualized on CXR.

  8. Previous resection lung surgery and history of lung tumor; 9. Cardiac pacemaker or implantable defibrillator

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males and females who were diagnosed with moderate-to-severe COPD by lung function studies and clinical evaluation
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2004-02; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Comparison of regional lung vibration energy with regional lung function
  To map regional lung vibration energy in patients with emphysema by using the lung image generated by the VRI system and compare findings to distibution of perfusion and ventilation in standard V/Q scans

SECONDARY OUTCOMES:
Correlation of vibration lung sound energy with regional lung functions by V/Q scan
  Evaluate if the regional vibration energy is correlated with regional lung functions, as assessed by V/Q scan

CONTACTS AND LOCATIONS:
Overall Officials: Issahar Ben-Dov, MD, Principal Investigator — Chaim Sheba Medical Center
Locations (1):
- Chaim Sheba Medical Center at Tel Hashomer, Ramat Gan, Israel

REFERENCES:
- [Background] Celli BR, MacNee W; ATS/ERS Task Force. Standards for the diagnosis and treatment of patients with COPD: a summary of the ATS/ERS position paper. Eur Respir J. 2004 Jun;23(6):932-46. doi: 10.1183/09031936.04.00014304. No abstract available. PMID 15219010
- [Background] Demir T, Ikitimur H, Akpinar Tekgunduz S, Mutlu B, Yildirim N, Akman C, Ozmen O, Kanmaz B. The relationship between pulmonary function tests, thorax HRCT, and quantitative ventilation-perfusion scintigraphy in chronic obstructive pulmonary disease. Tuberk Toraks. 2005;53(4):347-53. PMID 16456733
- [Background] Kramer MR, Raviv Y, Hardoff R, Shteinmatz A, Amital A, Shitrit D. Regional breath sound distribution analysis in single-lung transplant recipients. J Heart Lung Transplant. 2007 Nov;26(11):1149-54. doi: 10.1016/j.healun.2007.07.039. PMID 18022081
- [Background] Ikonen T, Harjula AL, Kinnula V, Savola J, Sovijarvi AR. Selective assessment of single-lung graft function with 133Xe radiospirometry in acute rejection and infection. Chest. 1996 Apr;109(4):879-84. doi: 10.1378/chest.109.4.879. PMID 8635364
- [Background] Guntupalli KK, Reddy RM, Loutfi RH, Alapat PM, Bandi VD, Hanania NA. Evaluation of obstructive lung disease with vibration response imaging. J Asthma. 2008 Dec;45(10):923-30. doi: 10.1080/02770900802395496. PMID 19085584